CLINICAL TRIAL: NCT06884189
Title: Pilot Study on the Exposure of Operators, Residents and Workers to Plant Protection Products Used in Apple Orchards and Possible Health Effects
Brief Title: Application of Plant Protection Products (PPP) in Apple Orchards
Acronym: aPPPle
Status: Recruiting | Type: Observational
Sponsor: German Federal Institute for Risk Assessment (Other)
Collaborators: Federal Ministry of Food and Agriculture (Unknown); ESTEBURG Obstbauzentrum Jork Kompetenzzentrum für den norddeutschen Obstbau (Unknown)
Responsible Party: Sponsor
Other Study IDs: 02
Record Dates: First submitted 2025-03-07; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Dermal Exposure; Inhalative Exposure; Metabolites in Urine; Effekt Biomarker in Blood
Keywords: exposure study; plant protection products; human biomonitoring; effect biomarker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Operators: People who apply plant protection products to apple crops.
- Workers: People who do manual work in apple cultivation, like pruning or harvesting.
- Residents: People whose place of residence is adjacent to the orchard under investigation.
- Control: People whose place of residence is at least 10 km away from agricultural apple orchards and a maximum of 150 km away from the apple orchard under investigation.

SUMMARY:
The aim of the aPPPle pilot study is to test feasibility and generate first results in preparation for a main study. The aPPPle study will investigate the exposure of operators, workers and residents to plant protection products (PPP) and potential physiological effects on blood biomarkers. The target plants are apple crops, as application occurs at higher altitudes and therefore higher drift/exposure is expected compared to ground-level application. The substances to be investigated are acetamiprid (an insecticide) and dithianon and dodine (two fungicides).

ELIGIBILITY:
Inclusion Criteria:

* belonging to one of the defined study groups
* over 18 years of age at the time of recruitment
* person can understand the language and content of the study requirements
* person is capable of consenting to participate in the study and has given written consent to participate in the aPPPle study
* person has health insurance

Exclusion Criteria for residents and control:

person has direct professional contact with the tested substances acetamiprid, dithianon or dodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Users, residents and workers:
  people from "Altes Land", a large apple-growing region in northern Germany
  Control: live at least 10 km and max. 150 km away from agricultural apple orchards
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Concentration of plant protection substances/metabolites in different matrices | Operators: during the observed work with PPP and for urine up to 48 hours after; resident: during the observed application and for urine up to 48 hours after; workers: during work in the orchards and for urine up to 48 hours a; control: at one time point
  The concentrations of the investigated substances/their metabolites will be analysed in urine, patches (to assess dermal exposure of the body), hand wipes (to assess dermal exposure of the hands), filters of an personal air sampler (to assess inhalation exposure), hair samples and gras samples
Effect biomarkers in blood and metabolome in plasma | enrollment until 7 days after application/work in the apple orchards; for people from the control group at one time point
  Defined effect biomarkers in blood as well as the metabolome in plasma will be analysed before and after application of plant protection products to observe possible early physiological changes.
  The following effect biomarkers in the blood will be measured:
  c-reactive protein, fasting glucose, HbA1c, cortisol, oxidized LDL, complete blood count, thyrotropin (TSH), free T3 (fT3), free T4 (fT4), gamma GT, GOT (ASAT), GPT (ALAT), bilirubin, cystatin C, urea

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Institute for Risk Assessment, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No